CLINICAL TRIAL: NCT04738071
Title: International Multicenter Patent foRamen OVale & strokE (IMPROVE) Registry
Acronym: IMPROVE
Status: Active, not recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-19-597
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Patent Foramen Ovale; Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Sex: Female and male patients
  Interventions: Device: PFO closure
- Age >60 years of age: Patients younger or oder than 6o years of age
  Interventions: Device: PFO closure
- World region: Patients from different world regions: North America, Europe, Asia, Latin America
  Interventions: Device: PFO closure
- Stroke vs. TIA: Index event: stroke vs. TIA
  Interventions: Device: PFO closure
- Neurocardiology Teams: Patients assessed by a neurocardiology team
  Interventions: Device: PFO closure

INTERVENTIONS:
Device: PFO closure — PFO closure after stroke or transient ischemic attack

SUMMARY:
Patent foramen ovale (PFO) is a prevalent cause of ischemic stroke and transient ischemic attack (TIA) in young patients. Its role as a cause of cerebrovascular events in the older population is more controversial because of other competing causes are more frequent in the elderly. Recent randomized controlled trials (RCTs) have shown that PFO closure is associated with a 59% relative risk reduction in the risk of recurrent ischemic stroke. As such, the number of PFO closure procedures are expected to increase substantially in the upcoming years. Real world data (RWD) informing on the medical management, the risk of stroke recurrence, incident atrial fibrillation, and other outcomes in stroke patients with PFO, with and without PFO closure, will become crucial for understanding how results from RCTs are translated into clinical practice globally.

The IMPROVE (International Multicenter Patent foRamen OVale & strokE) Registry is an observational, multicenter, international registry of men and women with an ischemic stroke or TIA. The aim is to enroll 8,800 patient-years at ≥50 sites in ≥20 countries.

The IMPROVE Registry will provide important information about the management and related outcomes of patients with ischemic stroke or TIA and PFO throughout different regions of the world and across a wide spectrum of healthcare systems.

ELIGIBILITY:
INCLUSION CRITERIA (all of the following criteria should be fulfilled)

* Age ≥18 years
* Ischemic stroke or TIA within 5 years and 1 year before inclusion in the registry. Patients with cerebrovascular events occurred within one year before the inclusion in the registry should be part of the prospective cohort.

  * Ischemic stroke is defined as:

    * focal neurological deficit of central origin lasting ≥24 hours -except for death within 24hrs- with or without imaging confirmation of cerebral infarction; or
    * focal neurological deficit of central origin lasting <24 hours with corresponding imaging evidence of cerebral infarction; or
    * focal neurological deficit of central origin lasting <24 hours in patients receiving IV thrombolysis or endovascular thrombectomy with or without imaging confirmation of cerebral infarction; or
    * non-focal encephalopathy lasting more than 24 hours -except for death within 24hrs- with imaging evidence of cerebral infarction; or
    * acute and permanent retinal ischemia of arterial origin.
  * TIA is defined as:

    * focal neurological deficit of central origin lasting <24 hours without corresponding imaging evidence of cerebral infarction in patients not receiving IV thrombolysis or endovascular thrombectomy.
* Confirmed patent foramen ovale.

EXCLUSION CRITERIA:

Exclusion Criteria

* Age <18 years
* Venous stroke
* Stroke mimics
* Patients with incomplete data at 12 months after the index ischemic stroke or TIA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The IMPROVE registry aims to include patients from Asia, Europe, Oceania, North America and Latin America. Academic, non-academic, urban and rural sites will be included. Principal investigators will be neurologists, since a confirmed diagnosis of ischemic stroke or TIA is mandatory before enrolment.
Sampling Method: Probability Sample
Enrollment: 3730 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
Recurrent stroke | Duration of follow-up (minimum of 3 months)
  Recurrent hemorrhagic or ischemic stroke

SECONDARY OUTCOMES:
Incident atrial fibrillation | Duration of follow-up (minimum of 3 months)
  New diagnosis of atrial fibrillation after the index date
Proportion of patients undergoing PFO closure | Within 12 months of the index diagnosis of PFO after the stroke or transient ischemic attack
  Proportion of patients undergoing PFO closure

OTHER OUTCOMES:
Recurrent stroke or death | Duration of follow-up (minimum of 3 months)
  Recurrent hemorrhagic or ischemic stroke, or death
Recurrent stroke or myocardial infarction | Duration of follow-up (minimum of 3 months)
  Recurrent hemorrhagic or ischemic stroke, or myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Luciano A Sposato, MD, MBA (PI), Principal Investigator — London Health Sciences Centre, Western University (London, ON. Canada); Antonio Arauz, MD (Co-Pi), Principal Investigator — National Institute of Neurology and Neurosurgery Manuel Velasco Suárez
Locations (1):
- Heart & Brain Lab, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request and after the Approval of Western University Ethics Review Board